CLINICAL TRIAL: NCT07155629
Title: Neoadjuvant Treatment vs Upfront Surgery for Left Sided Pancreatic Cancer (LEFT-PANC) - a Study Protocol for a Prospective Randomized Multicenter Trial
Brief Title: Neoadjuvant Treatment vs Upfront Surgery for Left-Sided Pancreatic Cancer
Acronym: LEFT-PANC
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Hanna Seppänen, Principal Investigator, Adjunct Professor, Pancreatic surgeon, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUS-LeftPanc-2025
Record Dates: First submitted 2025-08-25; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Pancreatic Cancer Resectable
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Gemcitabine; Oxaliplatin; Irinotecan; Leucovorin; Fluorouracil; Taxes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perioperative chemotherapy (Experimental): Patients who undergo surgical resection will receive adjuvant chemotherapy with 4 cycles (2 months) of FOLFIRINOX (oxaliplatin 85 mg/m2, irinotecan 180 mg/m2, leucovorin 400 mg/m2, and 5-fluorouracil (400 mg/m2 bolus then 2400 mg/m2 over 46 h)) OR 2 cycles (2 months) of Gemcitabine 1000 mg/m2 over 30 min at day 1, 8, 15 of each 28-day cycle and capecitabine 830 mg/m2 ×2 daily for 3 weeks and one week rest of each 28-day cycle. Regimen changes due to toxicity are allowed.
  After 2 and 4 months of NAT, response imaging (multiphased body CT) is assessed at a local pancreatic MDT. If stable disease or regression is observed, patients will undergo surgery after chemotherapy break of 3-6 weeks. Adjuvant chemotherapy (2-4 months) must be started within 4-12 weeks after resection. Dose adjustments follow local practice; adjuvant therapy depends on patient condition (mFOLFIRINOX, Gem+capecitabine, or gemcitabine alone).
  Interventions: Drug: mFOLFIRINOX neoadjuvant chemotherapy / Nab-paclitaxel and gemcitabine
- Control arm (No Intervention): After randomization, arm B patients are scheduled for upfront surgery. Adjuvant chemotherapy of 6 months must be started within 4-12 weeks after resection. Dose reduction or dose delays are acted upon according to local clinical practice at each centre. The adjuvant therapy is decided and if necessary modified according to patient's condition (mFOLFIRINOX, Gem+cabecitabine, single Gem).

INTERVENTIONS:
Drug: mFOLFIRINOX neoadjuvant chemotherapy / Nab-paclitaxel and gemcitabine — The benefits of neoadjuvant chemotherapy before surgery in a prospective multicenter randomized setting for resectable left-sided pancreatic cancer patients.
  Other Names: oxaliplatin; irinotecan; leucovorin; 5-fluorouracil; gemcitabine; Nanoparticle albumin bound paclitaxel
  Arms: Perioperative chemotherapy

SUMMARY:
Pancreatic cancer is one of the most treatment resistant malignancies, often diagnosed at a late stage and associated with poor survival. The 5-year overall survival rate remains around 10%. Prognosis is affected by multiple factors including tumor stage, biology, treatment response, and anatomical location. Distal (left-sided) pancreatic cancer, originating from the body or tail of the pancreas, accounts for approximately 20-25% of all pancreatic cancers and has been associated with worse survival than pancreatic head cancer, even when adjusted for stage. This may be due to histological, molecular, and embryological differences, and varied systemic therapy responses.

Neoadjuvant chemotherapy has become increasingly important in managing pancreatic cancer. It may improve outcomes by reducing tumor size, allowing for more complete (R0) resections, treating micrometastatic disease early, and identifying patients unlikely to benefit from surgery. While neoadjuvant therapy is recommended for borderline resectable and locally advanced tumors, randomized trials have not shown benefit for patients with upfront resectable pancreatic head cancer. Importantly, no randomized controlled trials have investigated the benefit of neoadjuvant treatment specifically in patients with upfront resectable left-sided pancreatic cancer, despite its distinct biology and worse prognosis.

Retrospective data suggest neoadjuvant therapy may improve survival in left-sided tumors. A recent multicenter study reported significantly longer overall survival in patients treated with neoadjuvant therapy compared to upfront surgery alone. However, prospective randomized data are lacking.

This multicenter randomized trial aims to assess whether patients with resectable left-sided pancreatic cancer benefit from neoadjuvant chemotherapy compared to upfront surgery. The study will reflect real-world clinical practice by allowing both commonly used regimens-FOLFIRINOX and Gemcitaine-Nab-paclitaxel -as neoadjuvant options. Previous studies have shown these regimens to be similarly effective, and switching between them due to toxicity or progression is feasible and does not seem to impair surgical outcomes or survival. This study aims to evaluate the benefits of neoadjuvant chemotherapy before surgery in a prospective multicenter randomized setting for resectable left-sided pancreatic cancer patients.

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized phase III trial evaluating whether neoadjuvant chemotherapy improves overall survival in patients with resectable left-sided (body/tail) pancreatic cancer compared to the current standard of upfront surgery followed by adjuvant chemotherapy.

Eligible patients have histologically confirmed pancreatic adenocarcinoma located in the body or tail of the pancreas, ECOG/WHO performance status 0-2, and radiologically resectable disease according to NCCN criteria. Patients are randomized 1:1 to receive either:

1. neoadjuvant chemotherapy, followed by surgery and adjuvant therapy, or
2. upfront surgery followed by adjuvant chemotherapy.

Randomization uses a minimization method with stratification by performance status, CA19-9 level, treatment center, and chemotherapy regimen. Surgery is scheduled within 4-6 weeks of randomization (control arm) or after the last neoadjuvant cycle (intervention arm). Left pancreatectomy (open or minimally invasive) with standard lymphadenectomy and splenectomy is performed with complications reported using Dindo/Clavien classification and ISGPS criteria. Radical antegrade posterior pancreatosplenectomy may be performed when needed to ensure clear margins. Tumor response to neoadjuvant therapy will be evaluated by standardized histopathological grading.

Patients are followed with laboratory tests and CT imaging at the completion of adjuvant therapy and every six months thereafter until disease recurrence or up to five years after surgery. Quality of life is assessed at baseline, pre-surgery (in the neoadjuvant arm), 4 weeks post-op, and during follow-up using the EORTC QLQ-C30 and PAN26 instruments. Patients are followed for recurrence and survival every 6 months for up to 5 years. Safety is monitored per CTCAE v5.0, with SAEs and SUSARs reported per regulatory guidelines. An independent DSMB will review safety data. Blood and tumor samples will be stored for future translational research.

The primary endpoint is overall survival. A total of 381 patients will be enrolled over 36 months. The trial is powered to detect a hazard ratio of 0.70 with 80% power and a 5% significance level, requiring 247 events (deaths). Analysis will follow the intention-to-treat principle using Kaplan-Meier, log-rank test, and Cox regression. Pre-specified subgroup analyses will assess factors such as age, performance status, CA19-9, and tumor characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Resectable left pancreatic cancer according to NCCN criteria
* Written and informed consent
* Age > 18y
* ECOG 0-2
* Fit for surgery
* Fit for neoadjuvant chemotherapy

Exclusion Criteria:

* ECOG > 2
* Histology other than ductal adenocarcinoma
* Unable to give written consent
* < 18y

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 381 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2030-08-31 (Estimated); Study Completion 2030-08-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From randomization until death or study completion, up to approximately 5 years.
  Overall survival of participants, defined as the time from randomization until death from any cause, analyzed in the intention-to-treat (ITT) population.

CONTACTS AND LOCATIONS:
Overall Officials: Hanna Seppänen, Adj. Prof., Pancreatic surgeon, Principal Investigator — Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Oulu University Hospital, Oulu